CLINICAL TRIAL: NCT01702948
Title: Understanding the Neurocircuitry of Nicotine Addiction Using Repetitive Transcranial Magnetic Stimulation (rTMS)
Brief Title: Studying Nicotine Addiction With Transcranial Magnetic Stimulation
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912479; 12-DA-N479
Record Dates: First submitted 2012-10-06; First posted 2012-10-10 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2017-10-03

CONDITIONS: Nicotine Dependence
Keywords: Functional Magnetic Resonance Imaging (fMRI); Nicotine; Repetitive TMS (rTMS); fMRI
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

- Nicotine addiction often makes it difficult to stop smoking. Researchers want to understand the areas of the brain that are important in nicotine addiction. They will use a type of brain stimulation called repetitive transcranial magnetic stimulation (rTMS) to look at part of the brain that may be involved in nicotine addiction. They will see how these areas affect brain function, thinking, and decision making. For this study, rTMS will first be tested on nonsmokers, then smokers will be recruited at a later time.

Objectives:

- To study areas of the brain involved in nicotine addiction.

Eligibility:

- Individuals at least 18 years of age who do not smoke.

Design:

* Participants will be screened with a physical exam and medical history. They will also provide a urine sample.
* There will be four study sessions. The first session will involve a magnetic resonance imaging (MRI) scan. The other three visits will involve rTMS and MRI scans.
* The first MRI scan will take a baseline picture of the brain. Participants will also practice the tasks for the other three sessions in a mock scanner.
* At the next three visits, participants will have rTMS and MRI scans. Two visits will involve rTMS; the other visit will involve mock rTMS with no actual magnetic stimulation. During the MRI scans, participants will perform tasks that involve decision making.

DETAILED DESCRIPTION:
Objective: To investigate the neurocircuitry cognitive and affective processing relevant to nicotine addiction using repetitive Transcranial Magnetic Stimulation (rTMS). Specifically, we will examine insula neurocircuitry using a unilateral H-coil to deliver rTMS to the Right dorsolateral prefrontal cortex (R DLPFC) and insula. We will examine the effect of various stimulation parameters on behavior as well as on task based activation and resting state functional connectivity (rsFC) during fMRI scanning.

Study population: Up to 60 healthy adults who are non-smokers will be enrolled to achieve 28 completers.

Design: Within subject design with each subject completing 4 sessions: rTMS at two different stimulation frequencies and 2 sham sessions.

Outcome measures: Behavior on a decision making task and task based and resting state blood oxygen level-dependent (BOLD) activation in neural circuits relevant to nicotine addiction during fMRI scanning.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males and females 18 - 55 years of age
  2. Able to give valid informed consent
  3. Right-handed
  4. If the subject is female, of childbearing potential, and sexually active, she agrees to use a medically acceptable contraception, and not become pregnant for the duration of the study. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. Female patients of childbearing potential who are or who anticipate the possibility of becoming sexually active with a male partner must use either: (1) contraceptive pill or intrauterine device (IUD) or depot hormonal preparation (ring, injection implant); and/or (2) a barrier method of contraception such as diaphragm, sponge with spermicide, or condom. Women who are not sexually active do not have to agree to use one of the acceptable contraception methods. Contraceptive measures will be reviewed with female subjects at each visit prior to the TMS session.

EXCLUSION CRITERIA:<TAB>

1. Personal or first-degree family history of any clinically defined neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness.
2. Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head that cannot be safely removed.
3. Current use, or use in the past 4 weeks of any investigational drug or of any medications with psychotropic, anti or pro-convulsive action
4. Increased intracranial pressure (lowers seizure threshold)
5. Lifetime history of major depressive disorder, schizophrenia, bipolar disorder, mania, or hypomania or current substance abuse or dependence or past dependence by DSM IV criteria, or urine toxicology positive for any illicit substance.
6. History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or any heart condition currently under medical care.
7. Pregnant or nursing women or women with reproductive potential who are sexually active and not using an acceptable form of contraception.
8. Any history of seizure

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2012-09-10; Study Completion 2017-10-03

PRIMARY OUTCOMES:
Behavior on a decision making task and task based and resting state BOLD activation in neural circuits relevant to nicotine addiction during fMRI scanning.

CONTACTS AND LOCATIONS:
Overall Officials: Mary R Lee, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Ahmed MA, Darwish ES, Khedr EM, El Serogy YM, Ali AM. Effects of low versus high frequencies of repetitive transcranial magnetic stimulation on cognitive function and cortical excitability in Alzheimer's dementia. J Neurol. 2012 Jan;259(1):83-92. doi: 10.1007/s00415-011-6128-4. Epub 2011 Jun 14. PMID 21671144
- [Background] Baeken C, De Raedt R, Van Schuerbeek P, Vanderhasselt MA, De Mey J, Bossuyt A, Luypaert R. Right prefrontal HF-rTMS attenuates right amygdala processing of negatively valenced emotional stimuli in healthy females. Behav Brain Res. 2010 Dec 25;214(2):450-5. doi: 10.1016/j.bbr.2010.06.029. Epub 2010 Jul 1. PMID 20600336
- [Background] Baumgartner T, Knoch D, Hotz P, Eisenegger C, Fehr E. Dorsolateral and ventromedial prefrontal cortex orchestrate normative choice. Nat Neurosci. 2011 Oct 2;14(11):1468-74. doi: 10.1038/nn.2933. PMID 21964488